CLINICAL TRIAL: NCT04075006
Title: Adjunct Low Dose Ketamine Infusion Versus Standard of Care in Mechanically Ventilated Critically Ill Patients at a Tertiary Saudi Hospital: Randomized, Prospective, Pilot Trial
Brief Title: Analgosedative adjuncT keTAmine Infusion iN Mechanically vENTilated ICU Patients
Acronym: ATTAINMENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Mohammed Bawazeer, Consultant Intensivist, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2191187; SCTR #19063002 (Other: Saudi Food and Drug Authority); ISRCTN14730035 (Registry Identifier: Current Controlled Trials)
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Critical Illness; Sedation; Mechanical Ventilation
Keywords: Ketamine, standard of care, critically ill, mechanically ventilation, ATTAINMENT, propofol, Fentanyl , midazolam , delirium, vasopressors
MeSH Terms: conditions — Critical Illness; Delirium | interventions — Ketamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Experimental): adjunct low dose continuous infusion ketamine in addition to the standard of care. Ketamine will be given at a fixed infusion rate of 0.12 mg/kg/hr (2 µg/kg/min) in the first 24 hours followed by 0.06 mg/kg/hr (1 µg/kg/min) in the second 24 hours, then discontinued
  Interventions: Drug: Ketamine
- Control Group (No Intervention): Standard of care in the ICU including propofol and / or fentanyl and/or midazolam according to KFSHRC sedation and analgesia protocol.

INTERVENTIONS:
Drug: Ketamine — standard of care plus Ketamine infusion at a fixed rate of 0.12 mg/kg/hr (2 µg/kg/min) in the first 24 hours followed by 0.06 mg/kg/hr (1 µg/kg/min) in the second 24 hours, then discontinued
  Arms: Ketamine Group

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of a low dose ketamine infusion used in combination of standard of care in critically ill patients to test whether ketamine can help to shorten the time of being in breathing tube and ventilator compared to the standard of care alone.

DETAILED DESCRIPTION:
Ketamine is used to produce sedation and relieve pain to minimize discomfort while a breathing tube placed in trachea (windpipe) and a machine (ventilator) used in the ICU. Several publications have shown that a low-dose ketamine in combination to opioids has been used to relieve acute pain after surgery. Ketamine has a favorable characteristics including bronchodilation, increase in blood pressure, does not cause constipation , maintain respiratory reflexes (respiratory spontaneous responses) make it an especially viable alternative for patients with unstable respiratory and hemodynamic function. However, the majority of these trials are conducted in a surgical ICU setting, retrospective in nature or randomized controlled clinical trials focusing on comparison of ketamine to placebo or two study drugs (e.g. ketamine versus opioid), despite the fact that most ICU patients are sedated with a combination of drugs. Moreover, the majority of those trials has a limited focus on patient-centered outcomes, as the primary outcome.

The aim of this study is to assess weather ketamine can help to shorten the time of being in breathing tube and ventilator (duration of mechanical ventilation). This is a prospective, randomized, active controlled, open-label pilot study to assess the efficacy and safety of Analgo-sedative adjuncT keTAmine Infusion iN Mechanically vENTilated ICU patients (ATTAINMENT trial). The study hypothesis is that low dose ketamine infusion will reduce the duration of mechanical ventilation with an acceptable safety profile compared to standard of care. The study will include adult ICU patients (> 14 years old) admitted to KFSHRC ICUs within the previous 24 hours, placed on the ventilator, expected to need breathing tube for longer than 24 hours and placed on KFSHRC sedation and pain protocol. Patients will be separated to 2 groups: The intervention group: will receive a low dose ketamine infusion used in combination of standard of care. Ketamine will be given as intravenous infusion at a fixed infusion rate 0.12 mg/kg/hr (2 µg/kg/min) in 1st 24hr followed by 0.06 mg/kg/hr (1 µg/kg/min) in 2nd 24hr. The control group which will receive standard of care in the ICU including propofol and / or fentanyl and/or midazolam according to KFSHRC ICU sedation and analgesia protocol as chosen by the treating clinician.The randomization process is computer-generated using block randomization with a size of 8 patients in each block.

The number of the subjects to be enrolled in this study is 80 and duration of the subject's participation is 48hrs. Patients will be assessed for duration of mechanical ventilation as a primary outcome.

Study medication (i.e. ketamine) will be administered until one the following occurs:

1. Patient has received ketamine for 48 hours (intended duration if the study), or
2. If ICU team deemed excessive sedation persisted after holding or decreasing the sedating medication and patient not on target sedation score called RASS,
3. Patient died or goal of care changed to comfort care
4. Patient extubated and sedation weaned off ,
5. an adverse event potentially attributable to the study drug is experienced by a patient that is deemed, in the opinion of the investigative team to warrant discontinuation of therapy such as fast heart beat persist >150 beat per min for more than 3 hours, high systolic blood pressure persist > 180 for more than 3 hours, severe agitation and pulling off breathing tube or lines, and aggressive behavior to the nursing staff.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ICU (Medical or surgical) patients (> 14 years old)
2. Mechanically ventilated within the previous 24 hours and expected to remain intubated for more than 24 hours.
3. The patient requires ongoing sedative medication
4. No objection from the ICU attending MD for enrollment

Exclusion Criteria:

1. Patients with a history of dementia or psychiatric disorders or on any anti-psychotics or anti-depressants medications at home
2. Pregnancy
3. Age < 14 years old
4. Expected to need mechanical ventilation less than 24 hours
5. Known hypersensitivity to ketamine
6. Patient on dexmedetomidine as primary sedative agent prior to randomization
7. Patients with cardiogenic shock, heart failure, myocardial infarction
8. History of end-stage liver disease.
9. Proven or suspected primary neurological injury (traumatic brain injury, ischemic stroke, intracranial hemorrhage, spinal cord injury, anoxic brain injury)
10. Patients with persistent heart rate (HR) > 150 bpm or systolic blood pressure (SBP) >180 mmHg
11. Patients who assigned as do-not-resuscitate order (DNR) or expected to die within 24 hours
12. Patients on ECMO
13. Patients with status epilepticus patients who are receiving the ketamine infusion for refractory status epilepticus
14. Proven or suspected status asthmaticus
15. Patients with expected targeted RASS of -5 such as patients on continuous infusion neuromuscular blockade

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Duration of Mechanical Ventilation | From Intubation to extubation date and off Mechanical Ventilation or until ICU discharge, death, or 28 days post randomization whichever occurs first.
  To assess whether ketamine can help to shorten the time of being in breathing tube and ventilator (duration of mechanical ventilation )

SECONDARY OUTCOMES:
Cumulative Sedation Dosages | First 48 hours after randomization
  To compare the cumulative dose of pain and sedative medications.
Dexmedetomidine use | First 48 hours after randomization
  To compare the number of patients started on dexmedetomidine.
Richmond Agitation Sedation Score (RASS) | First 48 hours after randomization
  To compare The number of patients are in RASS score goal.
Pain score | First 48 hours after randomization
  To compare The number of patients are in pain score goal. We will use the KFSHRC pain scale being used in our ICU.
  For Adult communicative patients, we will use a scale from 0-10. The "0" indicates "No pain" and "10" indicates "severe pain". Values between 1-3 indicate mild pain, values between 4-6 indicate moderate pain while values between 7-10 indicate severe pain.
  For non-communicative patients, A scale is composed of five categories: Physiology, Facial expressions, Activity (movement), Guarding And Respiratory, will be used. Each Category has a scale 0-2, then the total score is calculated and should be between 0-10. Values between 0-2 indicate no pain, values 3-6 indicate moderate pain while values between 7-10 indicate severe pain.
Vasopressor Medication Dosages | First 48 hours after randomization.
  To compare vasopressor requirement.
Hemodynamics | First 48 hours after randomization
  Changes in Mean Arterial Blood Pressure (MAP) and Heart Rate (HR)
Frequency of endotracheal tube Suctioning | First 48 hours after randomization
  Proportion of patient with changes in requirements of suctioning frequency to 2 hours of less
Hospital Length of Stay (LOS) | Throughout study completion (1 year)
  To compare hospital LOS
ICU Length of stay (LOS) | Throughout study completion (1 year)
  To compare ICU LOS
Tracheostomy | 28 days after randomization
  Tracheostomy rate
Unplanned extubation | 28 days after randomization
  Rate of unplanned extubation
Re-intubation rate | 28 days after randomization
  Rate of unplanned and unexpected re-intubation

OTHER OUTCOMES:
Incidence of Delirium | 48 hours after randomization
  Rate of positive Confusion Assessment Method in Intensive Care Unit (CAM-ICU)
The use of anti-psychotics | 48 hours after randomization
  Rate of using anti-psychotics for confirmed ICU-acquired delirium
Use of Physical restraints | 48 hours after randomization
  Use of physical restraints
Mortality | 28 days after randomization
  Death that occurs during 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Amer M, Maghrabi K, Bawazeer M, Alshaikh K, Shaban M, Rizwan M, Amin R, De Vol E, Baali M, Altewerki M, Bano M, Alkhaldi F, Alenazi S, Hijazi M. Adjunctive ketamine for sedation in critically ill mechanically ventilated patients: an active-controlled, pilot, feasibility clinical trial. J Intensive Care. 2021 Aug 30;9(1):54. doi: 10.1186/s40560-021-00569-1. PMID 34462007
- [Derived] Bawazeer M, Amer M, Maghrabi K, Alshaikh K, Amin R, Rizwan M, Shaban M, De Vol E, Hijazi M. Adjunct low-dose ketamine infusion vs standard of care in mechanically ventilated critically ill patients at a Tertiary Saudi Hospital (ATTAINMENT Trial): study protocol for a randomized, prospective, pilot, feasibility trial. Trials. 2020 Mar 20;21(1):288. doi: 10.1186/s13063-020-4216-4. PMID 32197636